CLINICAL TRIAL: NCT03196245
Title: NK Cell Mediated Influenza Immunity During Pregnancy
Acronym: Flu vaccine
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Doris Duke Charitable Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Catherine Blish, Assistant Professor, Stanford University
Other Study IDs: IRB-25182
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related; Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We have peripheral blood mononuclear cells and plasma from a small number of subjects banked for future assessment of immunologic function, as specified in our consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women undergoing influenza vaccination or acutely infected with influenza
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — There is no intervention. This is a purely observational study. We enrolled pregnant women as they received a vaccine as part of their regular medical care; we did not administer the vaccine. We also enrolled pregnant women acutely infected with influenza.

SUMMARY:
Pregnant women have increased morbidity and mortality due to infection with influenza. Changes in T cell function have been proposed as possible mechanisms for this finding. We believe that pregnancy induced changes in NK cell phenotype and function also impact influenza immunity. This study will compare the immune response of pregnant women and controls to TIV influenza vaccination as a surrogate for infection. In addition pregnant women with flu like illness will be enrolled to evaluate changes in immune response following influenza infection as compared to vaccination.

DETAILED DESCRIPTION:
We will enroll a cohort of 94 healthy pregnant women from the Lucille Packard Children's Hospital Obstetrics Clinic from 2012-2017.

Women will be enrolled during their 2nd and 3rd trimesters, a time of high risk of complications from influenza infection. All subjects will provide blood samples at day 0, then be immunized with TIV as part of their regular medical care, and will return for additional blood samples on approximately days 7 and 28.

In accordance with minimal risk guidelines in pregnant women, a total of 50 cc of blood will be drawn across all three visits (20 cc, 20 cc, and 10 cc respectively).

An additional blood draw of 20 cc will be performed approximately 6 weeks postpartum to coincide with the standard postpartum obstetrical follow up.

This is a purely observational study. There is no treatment or randomization. Influenza vaccination is the standard of care during pregnancy and will not be influenced by our study design. All subjects will receive standard prenatal care, and will have access to maternal fetal medicine experts.

Volunteers for the flu like illness arm will be those who present to the Stanford Hospital and Clinics with active flu-like symptoms. If the volunteer is interested in participating in the study, Dr. Blish's staff will complete the consent process and continue with study procedures. For hospitalized inpatients, the initial visit will be conducted onsite in the hospital room. For patients seen at the outpatient clinics, the initial visit will be conducted at the outpatient clinic or at the Clinical Translational Research Unit (CTRU) using respiratory infection precaution procedures.

Volunteers are encouraged to complete a second study visit. However, if returning for the Visit 2 is a reason why a volunteer is unwilling to participate in the study, the volunteer may complete only the first study visit and the follow-up phone call in order to enroll. Volunteers will be encouraged to receive influenza vaccination (if they have not already done so) through their primary care physician after the acute illness has subsided.

Study Visit 1 (Day 0) Enrollment/Baseline

* Potential participants will be provided with a verbal description of the study (purpose and study schedule and procedures). They then will be asked if they have any questions and allowed to read/sign the consent form. The consent form will be signed prior to the performance of any study procedures.
* Review study eligibility criteria and collect an abbreviated medical history and current concomitant medication use.
* Obtain vital signs (oral temperature, blood pressure, pulse, and respiratory rate), height and weight. Whenever possible, information will be obtained from existing clinic or hospital records.
* Record information about history of present illness.
* Collect blood volume sample in 3 10 ml green top tubes (maximum volume not to exceed 30 mL).
* Collect two nasopharyngeal flocked swab specimens(one specimen for the research laboratory and one specimen for the clinical virology laboratory diagnosis if not already collected by the hospital or the clinic staff).
* Provide Memory Aid for volunteer to record course of illness, ILI resolution date and serious adverse events occurring during the study period.

Visit 1A (phone call follow-up 7-10 days after Visit 1)

* Study personnel will contact the volunteer to remind participant to record any changes and course of their flu-like illness on the Memory Aid provided.
* Subsequent study visit will be scheduled.

Visit 2 (Day 28 ± 7 after Visit 1), PREFERRED, BUT OPTIONAL

* Review of medications and Memory Aid or new-onset medical conditions, influenza-like illness and SAEs.
* Obtain vital signs (oral temperature, blood pressure, pulse, and respiratory rate), and weight
* Collect blood sample (maximum volume not to exceed 20 mL): in two 10 ml green top tubes
* Collect two nasopharyngeal flocked swab specimens (both swabs to be sent to research laboratory).

Early Termination Visit:

If a volunteer is terminated from the study early, every effort should be made to perform the following procedures:

* Review current health status and note any changes since the last visit. Solicit information regarding SAEs and record all concomitant medications. Any ongoing related SAEs will be followed to resolution or until a stable chronic condition has been established. Volunteers will be encouraged to permit continued follow-up of SAEs if necessary
* Obtain remaining blood samples, if possible.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (18-42 years of age)
* Pregnant women planning to receive the TIV seasonal influenza vaccine or Pregnant women presenting with influenza like illness

Exclusion Criteria:

* Oral immunosuppressive agents (inhaled steroids OK)
* Serious chronic illness including autoimmune disease or chronic viral infections (eg, systemic lupus erythematosis,HIV, hepatitis B or C)
* Malignancy or blood dyscrasia
* Type I or II diabetes or morbid obesity (pre-pregnancy BMI>40)(gestational diabetes ok)
* Presence of fetal cardiac abnormalities
* Receipt of blood or blood products within the last year
* Prior receipt of current seasonal influenza vaccine for influenza vaccine arm
* History of egg allergy for influenza vaccine arm

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We enrolled only pregnant women.
Study Population: We enrolled a cohort of 94 healthy pregnant women from the Lucille Packard Children's Hospital Obstetrics Clinic from 2012-2016. Women will be enrolled during their 2nd and 3rd trimesters following administration of the TIV influenza vaccine which is the standard of care for pregnant women.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
NK cell function | 2 years
  We are assessing the NK cell repertoire and anti-influenza NK cell function

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
There will be no IPD shared with other researchers.

REFERENCES:
- [Background] Le Gars M, Seiler C, Kay AW, Bayless NL, Starosvetsky E, Moore L, Shen-Orr SS, Aziz N, Khatri P, Dekker CL, Swan GE, Davis MM, Holmes S, Blish CA. Pregnancy-Induced Alterations in NK Cell Phenotype and Function. Front Immunol. 2019 Oct 23;10:2469. doi: 10.3389/fimmu.2019.02469. eCollection 2019. PMID 31708922
- [Result] Le Gars M, Kay AW, Bayless NL, Aziz N, Dekker CL, Swan GE, Davis MM, Blish CA. Increased Proinflammatory Responses of Monocytes and Plasmacytoid Dendritic Cells to Influenza A Virus Infection During Pregnancy. J Infect Dis. 2016 Dec 1;214(11):1666-1671. doi: 10.1093/infdis/jiw448. Epub 2016 Sep 21. PMID 27655870
- [Result] Kay AW, Blish CA. Immunogenicity and Clinical Efficacy of Influenza Vaccination in Pregnancy. Front Immunol. 2015 Jun 4;6:289. doi: 10.3389/fimmu.2015.00289. eCollection 2015. PMID 26089824
- [Result] Kay AW, Bayless NL, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Blish CA. Pregnancy Does Not Attenuate the Antibody or Plasmablast Response to Inactivated Influenza Vaccine. J Infect Dis. 2015 Sep 15;212(6):861-70. doi: 10.1093/infdis/jiv138. Epub 2015 Mar 4. PMID 25740957
- [Result] Kay AW, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Holmes S, Blish CA. Enhanced natural killer-cell and T-cell responses to influenza A virus during pregnancy. Proc Natl Acad Sci U S A. 2014 Oct 7;111(40):14506-11. doi: 10.1073/pnas.1416569111. Epub 2014 Sep 22. PMID 25246558